CLINICAL TRIAL: NCT05659576
Title: Reducing Acute Upper Gastrointestinal Side-Effects of Thoracic Irradiation
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-307
Record Dates: First submitted 2022-12-13; First posted 2022-12-21 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Radiation Esophagitis
Keywords: Gastrointestinal; Sucralfate; Radiation Therapy; Thoracic cancer; 22-307
MeSH Terms: interventions — Sucralfate

STUDY DESIGN:
Intervention Model Description: This is a two-arm randomized study. There will be two separate randomizations in this study, one vs. two-stage consent and sucralfate vs. control.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- One Stage Consent (Active Comparator): Patient will sign one consent form.
  Interventions: Other: One consent
- Two Stage Consent (Experimental): Patient will sign two consent forms.
  Interventions: Other: Two consent
- Sucralfate (Experimental): During their RT course, patients randomized to the PS arm will receive a prescription for either: 1) sucralfate, 1 gram/10 mL oral suspension or 2) sucralfate 1 gram tablets.
  Interventions: Drug: Sucralfate
- Usual Care (Active Comparator): Standard supportive care by using opioids.
  Interventions: Other: Usual Care

INTERVENTIONS:
Drug: Sucralfate — 1. Sucralfate, 1 gram/10 mL oral suspension "By mouth, take 10 mL twice a day until RT completion, with one dose 30-60 minutes prior to their midday meal and the second dose prior to bedtime".May increase frequency up to 4 times per day, per physician discretion". Or
  2. Sucralfate 1 gram tablets By mouth, take one (1) tablet mixed in 15-30 mL warm water twice a day until RT completion, with one dose 30-60 minutes prior to their midday meal and the second dose prior to bedtime".
  The frequency of sucralfate can be adjusted at anytime at the treating physician's discretion after the patient has started it at twice a day, and the patient may discontinue sucralfate at anytime after RT completion, per physician discretion. May increase frequency up to 4 times per day, per physician discretion".
  Arms: Sucralfate
Other: Usual Care — Standard supportive care by using opioids.
  Arms: Usual Care
Other: One consent — Patient will sign one consent form.
  Arms: One Stage Consent
Other: Two consent — Patient will sign two consent forms.
  Arms: Two Stage Consent

SUMMARY:
The purpose of the study is to explore options for preventing and reducing symptoms of radiation esophagitis (RE). The researchers will also look what symptoms participants experience, and whether there are differences in weight loss in participants.

DETAILED DESCRIPTION:
Embedded Randomized Study to Assess Two-Stage Consent Design:

There will be two separate randomizations in this study, one vs. two-stage consent and sucralfate vs. control. The will first approach patients and explain that we are comparing different methods of informing patients about trials. If the patients do not wish to participate in the consent trial, participants will be approached for consent onto the therapeutic trial using the twostage research consent.

Patients who decline or who are not approached to take part in the randomized compression of consent methods based on physician discretion, may still take part in the randomized comparison of sucralfate vs. control (therapeutic trial).

ELIGIBILITY:
Inclusion Criteria:

* Patients being treated with thoracic irradiation with high-risk esophageal dose as determined below:

Esophageal dose:

* V50 ≥ 15% (25-35 once daily fractions) or 40 twice-daily [BID] fractions)
* V40 ≥ 15% (15-24 once daily fractions or 30 twice-daily [BID] fractions)
* V30 ≥ 15% (10-14 once daily fractions)

  * Age 18 years of age or older.

Exclusion Criteria:

* Known inability to take Sucralfate (tablet and/or suspension form), per physician discretion
* PEG tube
* Actively taking any opioid pain medications prior to radiation therapy
* History of an opioid use disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2022-12-13 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Accrual rate (Two-stage consent part) | 1 year
  Determine accrual rate of two-stage consent compared to standard onestage consent.
Reduce opioid use | 2 years
  as measured by documented opioid use within the past 24 hours in the EMR at time of final weekly status check

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Shin, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Cancer Center Basking Ridge (All Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (All Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (All Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk-Commack (All Protocol Activities ), Commack, New York
  - Memorial Sloan Kettering Westchester (All Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (All Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm